

## **Observational and Non-Interventional Study (ONIS) using Existing Data Protocol**

| BI Study Number: | 0205-0548 |
|---|---|
| Title: | Hospitalization, mortality rates and costs associated with chronic obstructive pulmonary disease (COPD) in Distrito Federal, Brazil, before and after the change in 2018 state COPD protocol version – Real-world data |
| NCT number: | NCT06053541 |
| Medicinal product: | Tiotropium bromide (SPIRIVA® RESPIMAT®) |
| Date | 28-May-2021 |
| Page 1 of 4 | |

## **DF COPD Study Protocol**

**Objective:** to investigate potential different patterns on chronic obstructive pulmonary disease (COPD) mortality, hospitalizations, ICU usage rates and costs after the COPD protocol change in Distrito Federal (DF), Brazil, in August 2018, with a substitution of tiotropium in soft mist inhaler to glycopyrronium in dry powder inhaler.

Methods: To analyze DATASUS, Brazilian Ministry of Health Public Database, data from patients ≥ 40 years old hospitalization and mortality rates due to COPD International Classification of Diseases (ICD) listed in the COPD DF Protocol 12 months before the protocol change (MAT 1) and 12 months after (MAT 2).

**Table 1:** ICD filters, per the DF COPD Protocol<sup>1</sup>:

| J41.0 | Simple chronic bronchitis |
|-------|--------------------------------------------|
| J41.1 | Mucopurulent chronic bronchitis |
| J41.8 | Mixed simple and mucopurulent chronic |
| | bronchitis |
| J42 | Unspecified chronic bronchitis |
| J43.1 | Panlobular emphysema |
| J43.2 | Centrilobular emphysema |
| J43.8 | Other emphysema |
| J43.9 | Emphysema, unspecified |
| J44.0 | Chronic obstructive pulmonary disease with |
| | acute lower respiratory infection |
| J44.1 | Chronic obstructive pulmonary disease with |
| | (acute) exacerbation |
| J44.8 | Other specified chronic obstructive |
| | pulmonary disease |
| J44.9 | Chronic obstructive pulmonary disease, |
| | unspecified |

On DATASUS, data on DF 40 years old or older population hospitalization and mortality rates filtered by the ICDs listed in Table 1 will be analyzed. The searches generate a LOG in order to ensure methodology. The data will be available on Microsoft Excel.

 Table 2: Information Available in the Hospital DataSUS Database (SIH).

| DATASUS_COLUMN | DATA | MEANING |
|---|---|---|
| UF_ZI | 530000 | STATE CODE |
| ANO_CMPT | 2013 | YEAR |
| MES_CMPT | 1 | MONTH |
| N_AIH | 5312100277187 | Authorization of Admission Number (13 Numbers) Unique |
| CEP | 71693046 | ZIP CODE PATIENT |
| MUNIC_RES | 530160 | CITY CODE PATIENT |
| NASC | 19970917 | BIRTHDAY PATIENT |
| SEXO | 3 | GENDER |
| UTI_MES_IN | 0 | UTI USE INDICATION |
| QT_DIARIAS | 0 | QTY OF DAYS IN HOSPITAL |
| PROC_SOLIC | 301050074 | REQUIRED PROCEDURE COD |
| PROC_REA | 301050074 | PROCEDURE EXECUTED NUMBER |
| VAL_SH | 570,9 | PROCEDURE VALUE (R\$) |
| VAL_SP | 153 | PROCEDURE WORKER VALUE (R\$) |
| VAL_TOT | 723,9 | TOTAL COST VALUE (R\$) |
| VAL_UTI | 0 | TOTAL COST ICU (R\$) |
| DT_INTER | 20121201 | ADMISSION DATA |
| DT_SAIDA | 20121231 | HOSPITAL DISCHARGE DATA |
| DIAG_PRINC | J448 | ICD CODE DIAGNOSTHIC OF ADMISSION |
| IDADE | 15 | AGE |
| DIAS_PERM | 30 | NUMBER OF DAYS IN HOSPITAL |
| MORTE | 0 | DEATH INDICATION |
| CNES | 2650355 | HOSPITAL NATIONAL CODE |

## The following outcomes will be analyzed:

- 1. Number of hospital admissions with and without ICU admissions
- 2. Hospital admission mortality with and without ICU admissions
- 3. Total costs associated with COPD hospitalizations
- 4. Infirmary beds (General and ICU beds)

The statistical analyses will be performed with Mann-Whitney test considering a p <0.05 for statistical significance, as the DATASUS generates unpaired data. The collected data will generate an observational, cross-sectional study in the cohort of adult hospitalized COPD patients.

## References

 Governo do Distrito Federal. Protocolo de Atenção à Saúde: TRATAMENTO MEDICAMENTOSO DA DOENÇA PULMONAR OBSTRUTIVA CRÔNICA ESTÁVEL. Available at: http://www.saude.df.gov.br/wp-conteudo/uploads/2020/09/Protocolo-DPOC-SES-DF.pdf Accessed on 19 Feb 2021.